CLINICAL TRIAL: NCT01662869
Title: A Randomized, Phase III, Multicenter, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of Onartuzumab (MetMAb) in Combination With 5-Fluorouracil, Folinic Acid, and Oxaliplatin (mFOLFOX6) in Patients With Metastatic HER2-Negative, MET-Positive Gastroesophageal Cancer
Brief Title: A Study of Onartuzumab in Combination With mFOLFOX6 in Participants With Metastatic HER2-Negative and MET-Positive Gastroesophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YO28322; 2012-001402-23 (EudraCT Number)
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Leucovorin; onartuzumab; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Onartuzumab+mFOLFOX6 (Experimental): Participants will receive onartuzumab 10 milligrams per kilogram (mg/kg) intravenous (IV) infusion + mFOLFOX6 (oxaliplatin, folinic acid, and 5-fluoruracil) regimen. Participants will receive a maximum of 12 cycles (each cycle is 14 days) of mFOLFOX6 with onartuzumab. Participants whose disease has not progressed after 12 cycles of mFOLFOX6 with onartuzumab will continue treatment with onartuzumab until disease progression, unacceptable toxicity, or death.
  Interventions: Drug: 5-Fluoruracil; Drug: Folinic acid; Drug: Onartuzumab; Drug: Oxaliplatin
- Placebo+mFOLFOX6 (Placebo Comparator): Participants will receive onartuzumab matching placebo + mFOLFOX6. Participants will receive a maximum of 12 cycles (each cycle is 14 days) of mFOLFOX6 with placebo. Participants whose disease has not progressed after 12 cycles of mFOLFOX6 with placebo will continue treatment with placebo until disease progression, unacceptable toxicity, or death.
  Interventions: Drug: 5-Fluoruracil; Drug: Folinic acid; Drug: Oxaliplatin; Drug: Placebo

INTERVENTIONS:
Drug: 5-Fluoruracil — Participants will receive 5-fluorouracil 400 milligrams per square meter (mg/m^2) IV bolus and then 2400 mg/m^2 as a continuous IV infusion over 46-48 hours on Day 1 of every cycle until disease progression or at the maximum of 12 cycles, whichever occurs first.
Drug: Folinic acid — Participants will receive folinic acid 400 mg/m^2 IV infusion over 2 hours on Day 1 of every cycle until disease progression or at the maximum of 12 cycles, whichever occurs first.
Drug: Onartuzumab — Participants will receive onartuzumab 10 mg/kg IV infusion on Day 1 of every cycle (each cycle = 14 days) until disease progression, unacceptable toxicity, or participant or physician decision to discontinue treatment.
  Other Names: MetMAb, RO5490258, PRO143966
  Arms: Onartuzumab+mFOLFOX6
Drug: Oxaliplatin — Participants will receive oxaliplatin 85 mg/m^2 IV infusion over 2 hours on Day 1 of every cycle until disease progression or at the maximum of 12 cycles, whichever occurs first.
Drug: Placebo — Participants will receive onartuzumab matching placebo on Day 1 of every cycle (each cycle = 14 days) until disease progression, unacceptable toxicity, or participant or physician decision to discontinue treatment.
  Arms: Placebo+mFOLFOX6

SUMMARY:
This randomized, multicenter, double-blind, placebo-controlled study will evaluate the efficacy and safety of onartuzumab (MetMAb) in combination with 5-fluorouracil, folinic Acid, and oxaliplatin (mFOLFOX6) in participants with metastatic human epidermal growth receptor (HER) 2-negative and MET-positive adenocarcinoma of the stomach or gastroesophageal junction. Participants will be randomized in a 1:1 ratio to receive either onartuzumab or placebo in combination with mFOLFOX6. Participants may continue to receive onartuzumab or placebo until disease progression, unacceptable toxicity, participant or physician decision to discontinue treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the stomach or gastroesophageal junction with inoperable, metastatic disease, not amenable to curative therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy greater than (>) 3 months
* Presence of tissue sample for IHC assay of MET receptor and HER2 status
* Tumor (primary or metastatic lesion) defined as MET-positive by IHC
* Measurable disease or non-measurable but evaluable disease, according to the RECIST v1.1; Participants with peritoneal disease would generally be regarded as having evaluable disease and allowed to enter the trial
* For women who are not postmenopausal or surgically sterile; agreement to use an adequate method of contraception (hormonal implant) during the treatment period and for at least 90 days after the last dose of onartuzumab/placebo and 6 months after the last dose of oxaliplatin
* For men: agreement to use a barrier method of contraception during the treatment period and for 90 days after the last dose of onartuzumab/placebo and 6 months after the last dose of oxaliplatin

Exclusion Criteria:

* HER2-positive tumor (primary tumor or metastasis)
* Previous chemotherapy for locally advanced or metastatic gastric carcinoma (adjuvant or neoadjuvant chemotherapy must be completed at least 6 months prior to randomization)
* Prior treatment with investigational drugs that target the human growth factor (HGF) or MET pathway
* History of another malignancy within the previous 5 years, except for appropriately treated and presumed cured carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage 1 uterine cancer, and localized prostate cancer
* Pregnancy or lactation
* Receipt of an investigational drug within 28 days prior to study start
* Clinically significant gastrointestinal abnormalities, apart from gastric cancer, including uncontrolled inflammatory gastrointestinal diseases
* Significant history of cardiac disease
* Significant vascular disease
* Serious active infection at the time of randomization, or other serious underlying medical conditions that would impair the ability of the participant to receive protocol treatment
* Infection with human immunodeficiency virus, hepatitis B, or hepatitis C
* Radiotherapy within 4 weeks before start of study treatment
* Major surgery within 4 weeks before start of study treatment, without complete recovery
* Any condition (psychological, geographical) that does not permit compliance with study and follow-up procedures
* Peripheral neuropathy
* Prior unanticipated severe reaction to fluoropyrimidine therapy
* Known sensitivity or contraindication to any component of study treatment
* Active gastrointestinal bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) in the MET Immunohistochemistry (IHC) 2+/3+ Participant Subgroup | Baseline until death (up to approximately 38 months overall)
OS in the Intent-To-Treat (ITT) Population | Baseline until death (up to approximately 38 months overall)

SECONDARY OUTCOMES:
Duration of Response, as Assessed by Investigator Using RECIST v1.1 | Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 6 weeks for 12 months and thereafter every 12 weeks up to approximately 38 months overall)
Percentage of Participants with a Tumor Response of CR or PR or Stable Disease (SD, Maintained for At Least 6 Months) as Determined by the Investigator Using RECIST v1.1 | Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 6 weeks for 12 months and thereafter every 12 weeks up to approximately 38 months overall)
Percentage of Participants with Adverse Events | Baseline up to approximately 38 months
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) of Onartuzumab | Pre-dose (within 1 hour before infusion start) on Day 1 of Cycles 1 and 4, (cycle length = 14 days), at study drug discontinuation visit (up to 38 months)
Change from Baseline in ATAs Level of Onartuzumab | Baseline (pre-dose [within 1 hour before infusion start] on Cycle 1 Day 1), pre-dose on Cycle 4 Day 1 (cycle length = 14 days), at study drug discontinuation visit (up to 38 months)
Minimum Serum Concentration of Onartuzumab (Cmin) | Pre-dose (within 1 hour before infusion start) on Day 1 of Cycles 1, 2 and 4, 30 minutes after end of infusion (duration of infusion = 60 minutes) on Cycle 1 Day 1 (cycle length = 14 days), at study drug discontinuation visit (up to 38 months)
Maximum Serum Concentration (Cmax) of Onartuzumab | Pre-dose (within 1 hour before infusion start) on Day 1 of Cycles 1, 2 and 4, 30 minutes after end of infusion (duration of infusion = 60 minutes) on Cycle 1 Day 1 (cycle length = 14 days), at study drug discontinuation visit (up to 38 months)
Progression-Free Survival (PFS), as Assessed by Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in MET IHC 2+/3+ Participant Subgroup | Baseline up to disease progression or death due to any cause, whichever occurs first (up to approximately 38 months overall)
PFS, as Assessed by Investigator Using RECIST v1.1 in ITT Population | Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 6 weeks for 12 months and thereafter every 12 weeks up to approximately 38 months overall)
Percentage of Participants with a Tumor Response of Complete Response (CR) or Partial Response (PR) as Determined by the Investigator Using RECIST v1.1 in MET IHC 2+/3+ Participant Subgroup | Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 6 weeks for 12 months and thereafter every 12 weeks up to approximately 38 months overall)
Percentage of Participants with a Tumor Response of CR or PR as Determined by the Investigator Using RECIST v1.1 in ITT Population | Baseline up to disease progression or death due to any cause, whichever occurs first (assessed every 6 weeks for 12 months and thereafter every 12 weeks up to approximately 38 months overall)
European Organization for Research and Treatment Cancer Quality of Life Questionnaire (EORTC QLQ) Core 30 (EORTC QLQ-C30) Score | Day 1 of each treatment cycle (cycle length = 14 days) up to approximately 38 months
EORTC QLQ-Gastric cancer Specific Quality of Life Questionnaire (EORTC QLQ-STOC22) Score | Day 1 of each treatment cycle (cycle length = 14 days) up to approximately 38 months
European Quality of Life-5 Dimensions (EQ-5D) Questionnaire Score | Day 1 of each treatment cycle (cycle length = 14 days) up to approximately 38 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (103):
- United States (14):
  - Los Angeles, California
  - Denver, Colorado
  - Fort Myers, Florida
  - St. Petersburg, Florida
  - Chicago, Illinois
  - Albany, New York
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Providence, Rhode Island
  - Nashville, Tennessee
  - Austin, Texas
  - Tyler, Texas
  - Vancouver, Washington
- Australia (6):
  - Port Macquarie, New South Wales
  - Sydney, New South Wales
  - Herston, Queensland
  - Box Hill, Victoria
  - East Bentleigh, Victoria
  - Nedlands, Western Australia
- Belgium (3):
  - Bruges
  - Leuven
  - Sint-Niklaas
- Canada (3):
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Czechia (2):
  - Brno
  - Olomouc
- France (9):
  - Angers
  - Avignon
  - Besançon
  - Brest
  - Clichy
  - Marseille
  - Paris
  - Saint-Herblain
  - Toulouse
- Germany (8):
  - Bochum
  - Essen
  - Hamburg
  - Leipzig
  - Ludwigsburg
  - Mannheim
  - Marburg
  - München
- Guatemala City, Guatemala
- Hong Kong, Hong Kong
- Israel (3):
  - Jerusalem
  - Ramat Gan
  - Tel Aviv
- Italy (7):
  - Catanzaro, Calabria
  - Udine, Friuli Venezia Giulia
  - Rome, Lazio
  - Milan, Lombardy
  - Turin, Piedmont
  - Florence, Tuscany
  - Prato, Tuscany
- Malaysia (2):
  - Sabah, Sabah
  - Kuala Lumpur
- Mexico (3):
  - Aguascalientes
  - Monterrey
  - Oaxaca City
- Panama City, Panama
- Poland (6):
  - Bydgoszcz
  - Gdansk
  - Krakow
  - Lublin
  - Rybnik
  - Warsaw
- Russia (5):
  - Ivanovo
  - Omsk
  - Ryazan
  - Samara
  - Tula
- Singapore, Singapore
- Seoul, South Korea
- Spain (5):
  - Elche, Alicante
  - Barcelona, Barcelona
  - Santander, Cantabria
  - Madrid, Madrid
  - Zaragoza, Zaragoza
- Switzerland (2):
  - Lucerne
  - Zurich
- Taiwan (4):
  - Changhua
  - Kaohisung
  - Taichung
  - Taipei
- Thailand (4):
  - Bangkok
  - Chiang Rai
  - Hat Yai
  - Lopburi
- Turkey (Türkiye) (6):
  - Antalya
  - Edirne
  - Erzurum
  - Malatya
  - Samsun
  - Sıhhiye, Ankara
- United Kingdom (6):
  - Bristol
  - Cardiff
  - London
  - Manchester
  - Southampton
  - Sutton

REFERENCES:
- [Derived] Shah MA, Bang YJ, Lordick F, Alsina M, Chen M, Hack SP, Bruey JM, Smith D, McCaffery I, Shames DS, Phan S, Cunningham D. Effect of Fluorouracil, Leucovorin, and Oxaliplatin With or Without Onartuzumab in HER2-Negative, MET-Positive Gastroesophageal Adenocarcinoma: The METGastric Randomized Clinical Trial. JAMA Oncol. 2017 May 1;3(5):620-627. doi: 10.1001/jamaoncol.2016.5580. PMID 27918764